CLINICAL TRIAL: NCT07285642
Title: Brain and Peripheral Muscle Oxygenation in Patients With Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: fNIRS&Exercise
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Copd
Keywords: COPD; FNIRS; Brain; Quadriceps femoris
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise; Breathing Exercises; Stroop Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Experimental)
  Interventions: Other: Aerobic Exercise (Treadmill Walking); Other: Resistance Exercise (Upper and Lower Limb Strength Training); Other: Breathing Exercises; Other: Cognitive Task (Stroop Task)
- Healthy Individuals (Experimental)
  Interventions: Other: Aerobic Exercise (Treadmill Walking); Other: Resistance Exercise (Upper and Lower Limb Strength Training); Other: Breathing Exercises; Other: Cognitive Task (Stroop Task)

INTERVENTIONS:
Other: Aerobic Exercise (Treadmill Walking) — Participants perform treadmill walking for 15 minutes at 60% of the heart rate reserve (HRR), following a 2-minute warm-up period. Exercise intensity is calculated individually using the Karvonen formula. Continuous oxygenation monitoring is conducted via fNIRS (prefrontal cortex) and NIRS (vastus lateralis).
Other: Resistance Exercise (Upper and Lower Limb Strength Training) — Participants perform resistance exercises for upper and lower limb major muscle groups using 60% of one-repetition maximum (1RM). Each exercise consists of 12 repetitions per set, repeated for 15 minutes with 10-second rest intervals between sets. Movements include shoulder flexion/abduction/extension, hip flexion/abduction/adduction/extension, knee extension, and squatting.
Other: Breathing Exercises — Participants perform controlled breathing exercises including diaphragmatic, chest, and lateral basal breathing techniques. Each pattern is executed in 10-repetition cycles, repeated for 15 minutes with 10-second rest intervals. All sessions begin with pursed-lip breathing instruction and are performed in a seated position.
Other: Cognitive Task (Stroop Task) — A computerized color-word interference test (PsychoPy software) is administered before and after the exercise session to evaluate executive function and attention. Performance is analyzed in relation to concurrent fNIRS measurements from the prefrontal cortex.

SUMMARY:
This interventional study aims to investigate the acute effects of different types of exercise on cerebral and peripheral muscle oxygenation in patients with chronic obstructive pulmonary disease (COPD). Functional near-infrared spectroscopy (fNIRS) and near-infrared spectroscopy (NIRS) will be used simultaneously to measure oxygenation changes in the prefrontal cortex and the vastus lateralis muscle during rest, Stroop task performance, the six-minute walk test, aerobic, strengthening, and breathing exercises.

The study will compare COPD patients and age- and sex-matched healthy controls to determine how brain and muscle oxygenation responses differ between groups and among exercise modalities. The findings are expected to guide the design of safe, individualized pulmonary rehabilitation programs that optimize oxygenation without compromising safety.

DETAILED DESCRIPTION:
Functional near-infrared spectroscopy (fNIRS) and near-infrared spectroscopy (NIRS) allow real-time, non-invasive assessment of tissue oxygenation. Although widely used in neurology and exercise physiology, their application in pulmonary diseases such as COPD remains limited.

This study is designed as a non-randomized controlled, multidisciplinary trial conducted at Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul. The research team includes specialists in physiotherapy and rehabilitation, pulmonology, and neuroscience.

Participants will undergo a single standardized pulmonary rehabilitation (PR) session comprising three exercise modalities:Aerobic training, Peripheral strengthening exercises and Breathing exercises.

Before and after exercise, participants will perform the Stroop cognitive task to evaluate executive function and its relationship with cerebral oxygenation. Continuous fNIRS and NIRS monitoring will occur at rest, during each exercise, and during recovery.

ELIGIBILITY:
Inclusion Criteria

* Age 40-70 years
* Diagnosis of moderate-to-severe COPD (GOLD stage II-III)
* Stable disease (no exacerbation in previous 4 weeks)
* BMI 18.5-24.9 kg/m²
* Manual muscle strength ≥ 4 (MRC scale)
* Ability to perform exercise tests safely
* Written informed consent

Exclusion Criteria

* Severe comorbid conditions (uncontrolled cardiac, neurological, or orthopedic disease)
* Need for high-flow oxygen therapy (>2 L/min)
* History of cerebrovascular disease or transient ischemic attack
* Musculoskeletal or dermatological conditions impairing NIRS measurement sites
* Restrictive lung disease, interstitial lung disease, or small-airway disease
* Participation in an exercise program within the last 12 months

Healthy Controls

* Age 40-70 years
* No acute or chronic disease
* Non-smoker
* BMI 18.5-24.9 kg/m²
* No musculoskeletal limitations

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral oxygenation during exercise | Day 1
  fNIRS device (Artinis Brite Lite, The Netherlands) with 8-channel prefrontal montage, sampling at 10 Hz. Data analyzed with MATLAB-based Homer3 and NIRS-KIT software.

SECONDARY OUTCOMES:
Change in peripheral muscle oxygenation | Day 1
  NIRS device (Moxy, Fortiori Design LLC, Minnesota, USA). Parameters analyzed include minimum, maximum, and mean SmO₂ and tHb.
Cognitive performance (reaction time, accuracy in Stroop task) | Pre-exercise (baseline) and immediately post-exercise (within 5 minutes after final exercise).
  Cognitive performance measured as reaction time (ms) and accuracy (%) during a computerized Stroop task performed before and after the exercise session. This reflects acute changes in executive function and attention related to cerebral oxygenation.
Six-Minute Walk Distance (6MWD) | Baseline
  Functional exercise capacity assessed using the standardized 6-minute walk test according to American Thoracic Society (ATS) guidelines. Distance covered is recorded in meters. Test repeated twice to minimize learning effect, and the better result is used for analysis.
Perceived Dyspnea (Modified Borg Scale) | Day 1
  Participant-reported dyspnea level evaluated before and after each exercise modality using the Modified Borg Scale (0-10).
Physical Activity Level (IPAQ-Short Form) | Baseline
  Self-reported physical activity level evaluated using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). Results expressed in MET-min/week.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No